CLINICAL TRIAL: NCT00729911
Title: Ablation vs. Amiodarone for Treatment of Atrial Fibrillation in Patients With Congestive Heart Failure and an Implanted ICD/CRTD
Brief Title: Ablation vs Amiodarone for Treatment of AFib in Patients With CHF and an ICD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Collaborators: Casa Sollievo della Sofferenza IRCCS (Other); Catholic University, Italy (Other); Southlake Regional Health Centre (Other); Stanford University (Other); University of Kansas (Other); The University of Texas Medical Branch, Galveston (Other); University of Foggia (Other); Sutter Health (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AATAC-AF
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure
Keywords: Atrial fibrillation Ablation
MeSH Terms: conditions — Heart Failure | interventions — Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AF ablation (Active Comparator): Subjects assigned to the catheter ablation strategy will undergo catheter based AF ablation. The goal of the procedure is to achieve isolation of all 4 pulmonary veins.
  Subjects assigned to receive Amiodarone will have the oral medication initiated in an clinic setting.
  Interventions: Procedure: Atrial Fibrillation ablation
- Amiodarone (Active Comparator): Amiodarone is taken orally on a daily basis.
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Procedure: Atrial Fibrillation ablation — Radio-frequency catheter ablation of atrial fibrillation
  Arms: AF ablation
Drug: Amiodarone — Taken orally on a daily basis.
  Arms: Amiodarone

SUMMARY:
1. To determine if catheter-based atrial fibrillation (AF) ablation is superior to Amiodarone treatment for symptomatic persistent/permanent AF in ICD/CRTD patients with an impaired left ventricular function.
2. Hypothesis: AF ablation is better than Amiodarone for subjects with symptomatic persistent or permanent AF and impaired LV function in terms of recurrence of AF, quality of life, 6-minute walk distance, EF and total number of hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an dual chamber ICD or CRTD (with an existing functional atrial lead) with remote monitoring capabilities and EF <= 40% within the last 3 months by echocardiogram, nuclear imaging, MRI or cardiac catheterization,
2. Persistent or chronic symptomatic AF resistant to anti-arrhythmic medication other than Amiodarone. Resistant defined as recurrent AF of greater than 5 minutes duration at least once per month.
3. Therapeutic anticoagulation for at least three weeks prior to initiation of therapy
4. Ability to complete 6 minute walk test.
5. Age >= 18 years old. (Females must be either post-menopausal >12 months, practicing a protocol-acceptable method of birth control [defined as injectable or implantable hormonal contraceptives, oral contraceptives, intrauterine device, diaphragm plus spermicide], or have had a hysterectomy, bilateral oophorectomy, or tubal ligation performed at least 6 months prior to enrollment).
6. All patients optimized on CHF medications including beta-blocker and ace-inhibitor or angiotensin-receptor blocker.
7. patients receiving low dose amiodarone- <200 mg for 2 or less months

Exclusion Criteria:

The exclusion criteria are:

1. Reversible causes of AF such as pericarditis, hyperthyroidism,
2. Presently with Valvular Heart disease requiring surgical intervention
3. Presently with coronary artery disease requiring surgical intervention
4. Early Post-operative AF (within three months of surgery)
5. Previous MAZE or left atrial instrumentation
6. Prolonged QT interval
7. Hypothyroidism
8. Liver Failure
9. Life expectancy <= 2 years
10. Social factors that would preclude follow up or make compliance difficult.
11. Contraindication to the use of anti-arrhythmic medications and/or coumadin and heparin
12. Enrollment in another investigational drug or device study.
13. Patients with severe pulmonary disease i.e. COPD or asthma
14. Documented intra-atrial thrombus, tumor, or another abnormality which precludes catheter introduction
15. Any ophthalmologic disorders (other than requiring glasses for vision correction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2008-10; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to Recurrence of AF lasting longer than 15 seconds | 1 year

SECONDARY OUTCOMES:
Change in distance walked in 6-minute walk test | 1 year
Total number of hospitalizations during the trial period for each group | 1 year
Change in MLHF Quality of Life during trial period | 1 year
Change in EF during trial period | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation; Luigi Di Biase, MD, PhD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation
Locations (1):
- Texas Cardiac Arrhythmia Research Foundation, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Di Biase L, Mohanty P, Mohanty S, Santangeli P, Trivedi C, Lakkireddy D, Reddy M, Jais P, Themistoclakis S, Dello Russo A, Casella M, Pelargonio G, Narducci ML, Schweikert R, Neuzil P, Sanchez J, Horton R, Beheiry S, Hongo R, Hao S, Rossillo A, Forleo G, Tondo C, Burkhardt JD, Haissaguerre M, Natale A. Ablation Versus Amiodarone for Treatment of Persistent Atrial Fibrillation in Patients With Congestive Heart Failure and an Implanted Device: Results From the AATAC Multicenter Randomized Trial. Circulation. 2016 Apr 26;133(17):1637-44. doi: 10.1161/CIRCULATIONAHA.115.019406. Epub 2016 Mar 30. PMID 27029350